CLINICAL TRIAL: NCT03306992
Title: A Phase III Randomized Study Comparing the Effects of a Personalized Exercise Program (PEP) Against No Intervention in Patients With Stage I-IIIa Primary Non-Small Cell Lung Cancer or Secondary Lung Cancer Undergoing Surgical Resection
Brief Title: Precision-exercise-prescription for Lung Cancer Patients Undergoing Surgery: The PEP Study
Acronym: PEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI104671; 5R01CA211705-05 (NIH)
Record Dates: First submitted 2017-09-29; First posted 2017-10-11 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Non Small Cell Lung Cancer; Secondary Lung Cancer
Keywords: Exercise
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Exercise Program (Experimental)
  Interventions: Behavioral: Personalized Exercise Program
- Standard of Care - No Exercise (No Intervention)

INTERVENTIONS:
Behavioral: Personalized Exercise Program — The PEP intervention involves a combination of home-based exercise as well as in-patient exercise. The exercise modes will include basic transfer and calisthenics mobility, aerobic and resistance exercises and will be performed in various postures (supine, sitting, standing and walking) with variable challenges (level walking, bending, inclines, steps and squatting).
  For patients randomized to the Intervention Group (Group 1), the PEP intervention will be personalized, implemented, and modified (based on the patients AM-PAC mobility stage) by a licensed physical therapist in face-to-face, virtual, or phone meetings (~30-40 minutes). An exercise education manual, specifically developed for this study, will be used by the physical therapist to educate the patients on all aspects of starting and maintaining the exercise intervention.
  Arms: Personalized Exercise Program

SUMMARY:
This is a Phase 3 study aimed at investigating the effects of a personalized exercise program (PEP) in NSCLC patients (stage I, II, IIIa) and secondary lung cancer patients undergoing surgical treatment at the University of Utah and comparing the intervention to the current standard of care (no exercise program).

DETAILED DESCRIPTION:
This is a Phase 3 study aimed at investigating the effects of a personalized exercise program (PEP) in NSCLC patients (stage I, II, IIIa) and secondary lung cancer patients undergoing surgical treatment at the University of Utah and comparing the intervention to the current standard of care (no exercise program).

Eligible patients will be randomized between two arms (1:1 ratio) prior to the surgery and will be followed for approximately 6 months post-surgery:

* An Intervention Arm (referred to in materials as Group 1) which features pre- and post-surgery PEP interventions.
* A Control Arm (referred to in materials as Group 2) which does not include a personalized exercise program (the standard of care). Patients randomized to the Control Arm will be given the opportunity to participate in a PEP-intervention session providing exercise counseling after the 6 month assessment and will receive a free activity tracker for their participation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Diagnosis of primary lung cancer stage I, II, or IIIa OR secondary lung cancer.
* Disease amenable to surgical resection in the opinion of the treating surgeon.
* Patients must be able to follow directions and complete questionnaires and exercise diaries in English.
* Patients must agree to be randomly assigned to either Intervention or Control Group.

Exclusion Criteria:

* Deemed ineligible for surgery by the enrolling physician
* Abnormalities on screening physical exam judged by study physicians or supervising physical therapist to contraindicate participation in exercise program compliance.
* Alcohol or drug abuse as judged by study physicians.
* Significant mental or emotional problems that would interfere with study participation will be assessed by the NCCN Distress Thermometer. Any value higher than 7 will trigger further intervention, but ultimately enrollment into the clinical trial will be determined by the enrolling physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in mobility performance at baseline, 2 months and 6 months | Done at baseline, 2 and 6 months
  Six Minute Walk (6MW) distance.
  The distance patients can walk indoors on a 25 meters level smooth-surfaced track over the course of 6 minutes will be measured at baseline as well as at the time of discharge and at the 2 and 6 months follow-up.

SECONDARY OUTCOMES:
Evaluate the change Short Physical Performance Battery (SPPB) score | Done at baseline, 2 and 6 months
  Short Physical Performance Battery (SPPB) test scores
  A secondary endpoint associated with the evaluation of improvement in physical performance is the result of the short physical performance battery test. The SPPB score (ranging from 1 to 12) will be obtained for each patient at the time points described above. Medians will be obtained and compared for each arm.
Compare results from PROMIS Questionnaire done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months | Done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months
  Results from PROMIS questionnaires.
Compare results from FACT-L (Functional Assessment of Cancer Therapy-Lung) Questionnaire done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months | Done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months
  Results from FACT-L (Functional Assessment of Cancer Therapy-Lung) questionnaire
Compare results from FACIT-F (Chronic Illness Fatigue Scale) Questionnaire done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months | Done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months
  Results from FACIT-F (Chronic Illness Fatigue Scale) questionnaire.
Compare results from PSQI (Pittsburgh Sleep Quality Index) Questionnaire done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months | Done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months
  Results from PSQI (Pittsburgh Sleep Quality Index) questionnaire.
Compare results from BREQ-3 (Behavioral Regulation in Exercise Questionnaire 3) Questionnaire done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months | Done at baseline, discharge (6-10 days after surgery on average), 2 and 6 months
  Results from BREQ-3 (Behavioral Regulation in Exercise Questionnaire 3) questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Ulrich CM, Himbert C, Barnes CA, Boucher KM, Daniels B, Bandera VM, Ligibel JA, Wetter DW, Hess R, Kim J, Lundberg K, Mitzman B, Marcus R, Finlayson SRG, LaStayo PC, Varghese TK Jr. Precision Exercise Effect on Fatigue and Function in Lung Cancer Surgery: A Randomized Clinical Trial. JAMA Surg. 2025 May 1;160(5):495-519. doi: 10.1001/jamasurg.2025.0130. PMID 40072448
- [Derived] Assmann ES, Ose J, Hathaway CA, Oswald LB, Hardikar S, Himbert C, Chellam V, Lin T, Daniels B, Kirchhoff AC, Gigic B, Grossman D, Tward J, Varghese TK Jr, Shibata D, Figueiredo JC, Toriola AT, Beck A, Scaife C, Barnes CA, Matsen C, Ma DS, Colman H, Hunt JP, Jones KB, Lee CJ, Larson M, Onega T, Akerley WL, Li CI, Grady WM, Schneider M, Dinkel A, Islam JY, Gonzalez BD, Otto AK, Penedo FJ, Siegel EM, Tworoger SS, Ulrich CM, Peoples AR. Risk factors and health behaviors associated with loneliness among cancer survivors during the COVID-19 pandemic. J Behav Med. 2024 Jun;47(3):405-421. doi: 10.1007/s10865-023-00465-z. Epub 2024 Feb 28. PMID 38418709
- [Derived] Ulrich CM, Himbert C, Boucher K, Wetter DW, Hess R, Kim J, Lundberg K, Ligibel JA, Barnes CA, Rushton B, Marcus R, Finlayson SRG, LaStayo PC, Varghese TK. Precision-Exercise-Prescription in patients with lung cancer undergoing surgery: rationale and design of the PEP study trial. BMJ Open. 2018 Dec 16;8(12):e024672. doi: 10.1136/bmjopen-2018-024672. PMID 30559162

DOCUMENTS (1):
  • Study Protocol (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT03306992/Prot_000.pdf